CLINICAL TRIAL: NCT02131311
Title: A Clinical Study of the Effectiveness and Safety of a Disposable Intra-vaginal Device for Stress Urinary Incontinence
Brief Title: A Clinical Study of the Effectiveness and Safety of a Disposable Intra-vaginal Device for Stress Urinary Incontinence (SUI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012118
Record Dates: First submitted 2014-05-02; First posted 2014-05-06 (Estimated); Results first posted 2016-03-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-02

CONDITIONS: Stress Urinary Incontinence (SUI)
Keywords: single use; disposable; pessary; stress urinary incontinence; sui
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pessary (Experimental): disposable, single-use pessary
  Interventions: Device: disposable, single-use pessary

INTERVENTIONS:
Device: disposable, single-use pessary

SUMMARY:
This study will evaluate the effectiveness of the pessary device by assessing reduction in urine leakage in approximately 80 women with SUI. Efficacy will be assessed by pad weight gain, frequency of stress urinary incontinence events, and a quality of life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* be female 18 years or older;
* provide written informed consent prior to study participation and receive a signed copy;
* be in generally good health as determined by the Investigator;
* have a ≥ 3 month history of experiencing SUI (self reported);
* be willing to use the pessary investigational device to control stress urinary incontinence;
* be willing to comply with study requirements and instructions;

Exclusion Criteria:

* pregnant, lactating or planning to become pregnant during the study;
* within 3 months post partum;
* intrauterine device (IUD) placement of less than 6 months;
* has self-reported difficulty emptying her bladder;
* a history of Toxic Shock Syndrome (TSS) or symptoms consistent with TSS;
* experience difficulty inserting or wearing an intra-vaginal device, including a tampon;
* vaginal surgery, perineal surgery, uterine surgery, or abortion (spontaneous or induced) within the past 3 months;
* has any Screening laboratory value outside the laboratory reference range considered clinically significant by the Investigator which could impact the safety of the subject or the outcome of the study;
* for any reason, the Investigator decides that the subject should not participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall Severance, MD, Principal Investigator — Radiant Research, Inc.
Locations (1):
- Study Center, Chandler, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 145 subjects entered the 2-week baseline phase and 55 subjects dropped before treatment
Period: Overall Study
Arm/Group | Pessary
Started | 90
Completed | 86
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population
Arm/Group | Pessary
Number analyzed (Participants) | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (11.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders for Pad Weight Gain or SUI Episodes
Time Frame: from the 14-day baseline period to the last 7 days of 14-day device usage period
Population: Intent-to-Treat (ITT) population. The "Number of Participants Analyzed" is the number subjects with available (non-missing) data in week 2
Measure: Number; unit: percentage of subjects
Arm/Group | Pessary
Number analyzed (Participants) | 87
percentage of subjects | 69

2. Secondary Outcome: Change in Stress Urinary Incontinence Episodes
Description: change from baseline as measured as reduction (improvement) in stress urinary incontinence episodes. Positive values are indicative of efficacious outcome.
Time Frame: from the 14-day baseline period to the last 7 days of 14-day device usage period
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: episodes/usage period
Arm/Group | Pessary
Number analyzed (Participants) | 88
episodes/usage period | 1.46 [0.38 to 2.81]

3. Secondary Outcome: Change in Pad Weight Gain
Description: change from baseline as measured as reduction (improvement) in pad weight gain. Positive values are indicative of efficacious outcome.
Time Frame: from the 14-day baseline period to the last 7 days of 14-day device usage period
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: grams/usage period
Arm/Group | Pessary
Number analyzed (Participants) | 87
grams/usage period | 5.7 [1.23 to 16.7]

4. Secondary Outcome: Change in Quality of Life as Measured by Incontinence Impact Questionnaire (IIQ-7)
Description: The IIQ-7 is based on 7 questions referring to areas which may have been influenced or changed by accidental urine loss and/or prolapse. These questions are assigned a value of, 0 = 'Not at all,' 1= 'Slightly,' 2 = 'Moderately,' or 3 'Greatly.' The IIQ-7 is scored by taking the average score of items and then multiplying the average by 33 1/3 to put scores on a scale from 0 to 100. A lower score is considered less impact to quality of life and a higher score reflects more impact to quality of life. In the same manner, a reduction in scores from baseline reflects improved quality of life.
Time Frame: baseline and end-of-treatment
Population: Intent-to-Treat (ITT) population. The "Number of Participants Analyzed" is the number subjects with available (non-missing) data at end of treatment
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Pessary
Number analyzed (Participants) | 86
units on a scale | 24 [5 to 47]

5. Secondary Outcome: Change in Stress Urinary Incontinence Episodes
Description: as for outcome 2
Time Frame: from the 14-day baseline period to the first 7 days of 14-day device usage period
Population: Intent-to-Treat (ITT) population. The "Number of Participants Analyzed" is the number subjects with available (non-missing) data in week 1
Measure: Median (Inter-Quartile Range); unit: number of episodes/usage period
Arm/Group | Pessary
Number analyzed (Participants) | 88
number of episodes/usage period | 1.3 [0.43 to 2.41]

6. Secondary Outcome: Change in Pad Weight Gain
Description: as for outcome 3
Time Frame: from the 14-day baseline period to the first 7 days of a 14-day device usage period
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: grams/usage period
Arm/Group | Pessary
Number analyzed (Participants) | 87
grams/usage period | 4.68 [1.27 to 18.5]

7. Secondary Outcome: Percentage of Responders for Pad Weight Gain or SUI Episodes
Time Frame: from the 14-day baseline period to the first 7 days of 14-day device usage period
Population: as for outcome 5
Measure: Number; unit: percentage of subjects
Arm/Group | Pessary
Number analyzed (Participants) | 88
percentage of subjects | 67

ADVERSE EVENTS:
Time Frame: two weeks
Description: All adverse events reported by the subject from study initiation [Visit 1 (Screening)] until study completion [Visit 3 (End-of-Treatment)] were recorded.
Arm/Group | Pessary
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 6/90
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pessary (N=90)
Diarrhea (Gastrointestinal disorders) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The STUDY SITE and PRINCIPAL INVESTIGATOR agree that all data, calculations, interpretations, opinions and recommendations regarding the STUDY (hereinafter referred to as "RESULTS") shall be the property of P&G. The STUDY SITE and PRINCIPAL INVESTIGATOR agree to consider the RESULTS as INFORMATION subject to confidentiality restrictions